CLINICAL TRIAL: NCT03287193
Title: Identification of the Molecular and/or Pathophysiological Bases of Rare Diseases of Genetic Origin (or Rare Forms of Frequent Diseases Suspected of Being of Genetic Origin).
Acronym: DISCOVERY
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: OLIVIER-FAIVRE 2016
Record Dates: First submitted 2017-08-22; First posted 2017-09-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Rare Diseases of Genetic Origin; Rare Forms of Common Diseases Suspected of Being Genetic in Origin
MeSH Terms: interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood and/or tissue sampling — for patient and related person
Genetic: high-throughput sequencing — exome or whole genome sequencing

SUMMARY:
Rare diseases are conditions affecting a small number of people, requiring specific and often multidisciplinary medical care. There are over 7,000 rare diseases, around 80% of which are genetic in origin. These diseases are generally severe, chronic and progressive, and can considerably affect the quality of life of sufferers.

Although significant efforts in the search for genetic causes over the last two decades have led to the identification of thousands of genes associated with Mendelian diseases, half of all individuals with a rare disease remain without a genetic diagnosis. It is important to pursue the ambition of participating in the effort set by Europe, namely the identification of a large majority of the genetic causes responsible for rare diseases, and to be able to provide genetic counselling to patients and their families. In the past, scientific research to discover genes required a large number of families and individuals, and was long and costly to carry out. Today, this approach is facilitated by next-generation sequencing.

When high-throughput sequencing (HTS) identifies candidate genes or genetic abnormalities, it may be necessary to propose functional analyses to try to reach a conclusion.

ELIGIBILITY:
Inclusion Criteria:

-Patients (children or adults) with a suspected rare disease (or rare form of a common disease) of genetic origin for which the molecular basis is not known, or for which the understanding of the physiopathological mechanism is imperfectly known.

OR

-Foetuses with developmental abnormalities for which the molecular basis is not known, or for which the understanding of the physiopathological mechanism is imperfectly known.

OR

* Apparently healthy relatives or controls AND
* Consent of the patient or his/her legal representative
* Suitable level of understanding

Exclusion Criteria:

* Patients without national health insurance cover

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed at the Centre de Référence Anomalies du Développement du CHU de Dijon
Sampling Method: Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2017-03-13 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of new genes or genetic abnormalities identified. | through study completion, an average of 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France